CLINICAL TRIAL: NCT04148742
Title: A Phase I/II, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of DZD9008 in Patients With Non-Hodgkin B-cell Lymphoma
Brief Title: Assessing an Oral Bruton Tyrosine Kinase Inhibitor, DZD9008 in Patients Who Have Non-Hodgkin B-cell Lymphoma (WU-KONG3)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical development strategy adjustment, non-safety reason
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZ2019B0001
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Non-Hodgkin's B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- daily dose of DZD9008 (Experimental): daily dose of DZD9008
  Interventions: Drug: DZD9008

INTERVENTIONS:
Drug: DZD9008 — Daily dose of DZD9008, except for cycle 0 of Part A, in which a single dose of DZD9008 is administrated. Starting dose of DZD9008 is 50 mg once daily. If tolerated, subsequent cohorts will test increasing doses of DZD9008.

SUMMARY:
This study will treat patients with non-Hodgkin B-cell lymphoma who have relapsed from, refractory or intolerant to prior therapy. This study will help understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body and preliminarily assess its anti-cancer activity as monotherapy.

DETAILED DESCRIPTION:
A Phase I/II, Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of DZD9008 in Patients with Non-Hodgkin B-cell Lymphoma. This study includes dose escalation (Part A) and dose expansion (Part B).

ELIGIBILITY:
Inclusion criteria:

* Aged at least 18 years old.
* Patients must be willing and able to participate in all required evaluations and procedures.
* Patients must be able to provide a signed written informed consent.
* With documented histologically confirmed diagnosis of CLL/SLL, MCL or MZL and have least 1 measurable site of disease. Subjects must have relapsed, or are refractory or intolerant to >= 2 lines of prior therapy, and without preferred alternative treatment as judged by investigator. For Part B, subjects should be either BTK inhibitor treatment naive or intolerant to prior BTK inhibitor within 6 months on treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Predicted life expectancy ≥ 12 weeks.
* Adequate organ system functions.

Exclusion criteria:

* Prior malignancy requires active treatment within 2 to 3 years.
* A life-threatening illness, medical condition or organ system dysfunction.
* Radiotherapy with a limited field of radiation for palliation within 1 week of the screening.
* Major surgery within 4 weeks before screening.
* Prior treatment with any onco-immunotherapy within 4 weeks before screening.
* Subjects require immediate cytoreduction.
* Any history of Richter's transformation.
* Central nervous system (CNS) involvement unless previous treated and asymptomatic.
* Requires anticoagulation therapy with Warfarin, heparin.
* Known history of human immunodeficiency virus (HIV); Positive Hepatitis B surface antigen (HbsAg) or positive HCV antibodies; any other uncontrolled active systemic infection.
* Any of the following cardiac criteria: (1) mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs). (2) prior history of atrial fibrillation. (3) any factors that increase the risk of QTcF prolongation, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
* History of stroke or intracranial haemorrhage.
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection.
* History of hypersensitivity.
* Receiving (or unable to stop using) medications or herbal supplements known to be potent inhibitors or inducers of CYP3A.
* Grapefruit, grapefruit juice, and orange marmalade (made with Seville oranges) should be excluded.
* Women who are pregnant or breast feeding
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Previous allogenic bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of Treatment-Emergent Adverse Events | Through study completion, an average of 1.5 years
  Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE v5.0
Part B: objective response rate (ORR) | Through study completion, an average of 1.5 years

SECONDARY OUTCOMES:
Maximum Plasma DZD9008 concentration | up to 16 weeks
Plasma DZD9008 concentration- Area Under the Curve | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Nanjing
  - Jiangsu Province Hospital - Haematology, Nanjing

IPD SHARING:
Plan to Share IPD: No